CLINICAL TRIAL: NCT05534048
Title: A Phase III Study to Evaluate the Safety and Immunogenicity of PTX-COVID19-B Administered as Booster Vaccination in Previously Vaccinated Adults Aged 18 Years and Older
Brief Title: Booster Study of PTX-COVID19-B in Adults Aged 18 Years and Older
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Everest Medicines (Singapore) Pte. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COVI-EM-002
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — PTX-COVID19-B COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Efficacy cohort and safety cohort are parallel conducted.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTX-COVID19-B (Experimental)
  Interventions: Biological: PTX-COVID19-B
- Comirnaty® (Active Comparator)
  Interventions: Biological: Comirnaty®

INTERVENTIONS:
Biological: PTX-COVID19-B — The vaccine product, PTX-COVID19-B, is a preservative-free, sterile mRNA-lipid nanoparticle (mRNA-LNP) dispersion in an aqueous cryoprotectant buffer intended for IM injection.
  Arms: PTX-COVID19-B
Biological: Comirnaty® — 0.45 mL concentrate in a 2 mL clear multidose vial (type I glass) with a stopper (synthetic Bromo-butyl rubber) and a purple flip-off plastic cap with aluminum seal. Each vial contains 6 doses.
  Arms: Comirnaty®

SUMMARY:
The purpose of this clinical trial is to Evaluate the Safety and Immunogenicity of PTX-COVID19-B Administered as Booster Vaccination in Previously Vaccinated Adults Aged 18 Years and Older.

This study is seeking participants who are:

Adult males and females 18 years of age or older; In efficacy cohort : Subjects who were previously vaccinated with 2 doses of Comirnaty® administered at least 3 months prior to the booster dose..

All participants in this efficacy cohort will receive 1 of the 2 study vaccines: PTX-COVID19-B or Comirnaty®.

All participants in efficacy cohort will receive a single 40 microgram dose PTX-COVID19-B of the study vaccine or one dose of Comirnaty® at the first study clinic and will return to the study clinic 6 more times. At each clinic visit, a blood sample will be taken. They study is about 6 months long for each participant.

In safety cohort: Subjects who have previously received any primary series approved by WHO Emergency Use Authorization at least 3 months prior to enrollment or subjects who have already received one authorized booster vaccination and planned to receive PTX-COVID19-B as the 4th shot will be enrolled.

All participants in this safety cohort will receive 1 dose vaccines: PTX-COVID19-B.

All participants in safety cohort will receive a single 40 microgram dose of the study vaccine at the first study clinic and will return to the study clinic 5 more times. At each clinic visit, a blood sample will be taken. They study is about 6 months long for each participant.

ELIGIBILITY:
Inclusion Criteria:

-

Efficacy Cohort:

Each subject must meet all of the following criteria to be enrolled into the Efficacy Cohort:

1. Subject is able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Adult males and females 18 years of age or older on the day of signing the ICF (or the legal age of consent in the jurisdiction in which the study is taking place)
3. Had document of previous primary vaccination of 2 doses of Comirnaty® at least 3 months on the day of signing the ICF
4. SARS-CoV-2 Reverse transcription-polymerase chain reaction (RT-PCR)-negative at screening.
5. Body mass index of ≥ 18 and ≤ 30 kg/m2 at screening.
6. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception (i.e., including hysterectomy, bilateral salpingectomy, and bilateral oophorectomy, hormonal oral [in combination with male condoms with spermicide], transdermal, implant, or injection, barrier [i.e., condom, diaphragm with spermicide]; intrauterine device; vasectomized partner [6 months minimum], clinically sterile partner; or abstinence) during the study or 6 months after the last study vaccine, whichever later.

   * A female subject is considered a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile.
   * Subjects not of childbearing potential are not required to use any other forms of contraception during the study. Non-childbearing potential is defined as subject confirmed: i. Surgical sterilization (e.g., bilateral oophorectomy, bilateral salpingectomy, bilateral occlusion by cautery [Essure System® is not acceptable], hysterectomy, or tubal ligation).

   ii. Postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to screening); if postmenopausal status is unclear, pregnancy tests will be performed prior to vaccinations.
7. WOCBP must have a negative pregnancy test before vaccination. If menopausal status is unclear, a pregnancy test is required.

Safety Cohort:

Each subject must meet all of the following criteria to be enrolled into the Safety Cohort:

1. Subject is able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Adult males and females 18 years of age or older on the day of signing the ICF (or the legal age of consent in the jurisdiction in which the study is taking place) in general good health before study participation with no clinically relevant abnormalities (at Investigator's discretion) that could interfere with study assessments. Subjects may have stable comorbidities (no change in medications, exacerbations, or hospitalizations in the past 3 months).
3. Have previously received any full primary series approved by WHO Emergency Use Authorization at least 3 months prior to enrollment or who have already received one authorized booster vaccination and planned to receive PTX-COVID19-B as the 4th shot.
4. SARS-CoV-2 Reverse transcription-polymerase chain reaction (RT-PCR)-negative at screening.
5. Body mass index of ≥ 18 and ≤ 30 kg/m2 at screening.
6. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception (i.e., including hysterectomy, bilateral salpingectomy, and bilateral oophorectomy, hormonal oral [in combination with male condoms with spermicide], transdermal, implant, or injection, barrier [i.e., condom, diaphragm with spermicide]; intrauterine device; vasectomized partner [6 months minimum], clinically sterile partner; or abstinence) during the study or 6 months after the last study vaccine, whichever later.

   * A female subject is considered a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile.
   * Subjects not of childbearing potential are not required to use any other forms of contraception during the study. Non-childbearing potential is defined as subject confirmed: i. Surgical sterilization (e.g., bilateral oophorectomy, bilateral salpingectomy, bilateral occlusion by cautery [Essure System® is not acceptable], hysterectomy, or tubal ligation).

   ii. Postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to screening); if postmenopausal status is unclear, pregnancy tests will be performed prior to vaccinations.
7. WOCBP must have a negative pregnancy test before vaccination. If menopausal status is unclear, a pregnancy test is required.

Exclusion Criteria:

-

Efficacy Cohort:

Subjects will not be eligible for Efficacy Cohort participation if they meet any of the exclusion criteria:

1. Individuals who are antigen positive, seropositive or reverse transcriptase polymerase chain reaction (RT-PCR) positive for SARS-CoV-2.
2. Women currently pregnant, lactating, or planning a pregnancy within 3 months post boost vaccine.
3. Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination including known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV);
4. Receipt of an organ or bone marrow transplant; or Long-term (>2 weeks) use of oral or parenteral steroids or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) within 6 months before screening (nasal and topical steroids are allowed).
5. History of Guillain-Barré Syndrome or any degenerative neurology disorder, or myocarditis, pericarditis.
6. History of anaphylactic-type reaction to any injected vaccines; or known or suspected hypersensitivity to 1 or more of the components of the vaccine.
7. Acute illness or fever (axillary temperature ≥ 37.5ºC or oral temperature ≥ 38.0ºC) within 3 days (72 hours) before study enrollment (enrollment may be delayed for full recovery if acceptable to the investigator).
8. Congenital or functional absence of spleen, complete or partial removal of spleen in any case.
9. Donate or loss ≥ 450 ml of blood within 1 month prior to enrollment or expected blood donation during the study.
10. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month (3 months for immunoglobulins) before enrollment in this study; or who expect to receive another experimental agent during participation in this study.
11. Receipt of immunoglobulin or another blood product within the 3 months before enrollment in this study or those who expect to receive immunoglobulin or another blood product during this study.
12. Ineligible for the study based on the assessment of investigator.
13. Suspected or known current alcohol or drug dependency within 12 months of screening.
14. Individuals who are using medications with the intention of COVID-19 prophylaxis and who received or voluntarily plan to receive any other COVID-19 booster vaccine other than the study vaccines.
15. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
16. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 30 days prior to first study vaccination.
17. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
18. Bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
19. Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e., warfarin) or novel oral anticoagulants (i.e., apixaban, rivaroxaban, dabigatran and edoxaban)
20. History of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2) or cerebral venous sinus thrombosis, increased risk for cerebrovascular venous and sinus thrombosis, history of immune thrombocytopenia, or a history of capillary leak syndrome.

Safety Cohort:

Subjects will not be eligible for Safety Cohort participation if they meet any of the exclusion criteria:

1. Individuals who are antigen positive or reverse transcriptase polymerase chain reaction (RTPCR) positive for SARS-CoV-2.
2. Subjects who have vaccinated with 2 or more booster shots and plan to receive PTXCOVID19-B as the 5th or more shot.
3. Women currently pregnant, lactating, or planning a pregnancy within 3 months post boost vaccine.
4. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
5. Receipt of an organ or bone marrow transplant; or Long-term (>2 weeks) use of oral or parenteral steroids or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) within 6 months before screening (nasal and topical steroids are allowed).
6. History of Guillain-Barré Syndrome or any degenerative neurology disorder, or myocarditis, pericarditis.
7. History of anaphylactic-type reaction to any injected vaccines; or known or suspected hypersensitivity to 1 or more of the components of the vaccine.
8. Acute illness or fever (axillary temperature ≥ 37.5ºC or oral temperature ≥ 38.0ºC) within 3 days (72 hours) before study enrollment (enrollment may be delayed for full recovery if acceptable to the investigator).
9. Congenital or functional absence of spleen, complete or partial removal of spleen in any case.
10. Donate or loss ≥ 450 ml of blood within 1 month prior to enrollment or expected blood donation during the study.
11. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month (3 months for immunoglobulins) before enrollment in this study; or who expect to receive another experimental agent during participation in this study.
12. Receipt of immunoglobulin or another blood product within the 3 months before enrollment in this study or those who expect to receive immunoglobulin or another blood product during this study.
13. Ineligible for the study based on the assessment of investigator.
14. Suspected or known current alcohol or drug dependency within 12 months of screening.
15. Individuals who are using medications with the intention of COVID-19 prophylaxis and who voluntarily plan to receive any other COVID-19 booster vaccine other than the study vaccines.
16. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
17. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 30 days prior to first study vaccination.
18. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
19. Bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
20. Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e., warfarin) or novel oral anticoagulants (i.e., apixaban, rivaroxaban, dabigatran and edoxaban)
21. History of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2) or cerebral venous sinus thrombosis, increased risk for cerebrovascular venous and sinus thrombosis, history of immune thrombocytopenia, or a history of capillary leak syndrome. syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3800 (Estimated)
Dates: Start 2023-02-03 (Estimated); Primary Completion 2023-07-02 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that the immune response of a single booster dose of PTX-COVID19-B is non inferior to that of Comirnaty® | Day15
  The 50% neutralizing antibody titers (NT50), as measured by pseudovirusbased neutralization assay (PBNA), at Day 15
To assess safety of booster vaccination of PTX-COVID19-B in Safety Cohort | Incidence of solicited AEs Day1-Day8; Incidence of unsolicited AEs Day1-Day29; Incidence of SAEs, MAAEs, NOCD, AESI, and PIMMC Day1-Day181
  * Incidence of solicited AEs;
  * Incidence of unsolicited AEs;
  * Incidence of SAEs, MAAEs, NOCD, AESI, and PIMMC

IPD SHARING:
Plan to Share IPD: Undecided